CLINICAL TRIAL: NCT00114920
Title: A Three-Stage, Modified-Blind, Dose-Escalating Study to Assess Efficacy and Safety of Resiquimod Gel for the Treatment of Common Warts in Adults
Brief Title: Twelve Week Safety and Efficacy Study With a Topical Gel to Treat Common Warts in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1508-RESI
Record Dates: First submitted 2005-06-20; First posted 2005-06-21 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2006-11

CONDITIONS: Warts
Keywords: Wart(s); Adults; Common Wart(s)
MeSH Terms: conditions — Warts | interventions — resiquimod

INTERVENTIONS:
Drug: Resiquimod

SUMMARY:
The primary purpose of this study is to evaluate the effectiveness in adults, of four different strengths of resiquimod gel applied to common wart(s) three times a week for twelve weeks.

A second purpose is to evaluate the safety of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of common warts
* Two forms of birth control

Exclusion Criteria:

* Pregnant or breast feeding
* Other types of wart(s), ie. plantar
* Currently participating in another clinical study
* Chronic viral hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2004-03

PRIMARY OUTCOMES:
Clearance of treated common wart(s)

SECONDARY OUTCOMES:
Partial clearance of treated common wart(s)
Wart recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Welborn Clinic, Evansville, Indiana, United States